CLINICAL TRIAL: NCT04263714
Title: Effect of Exercise on the Human Skeletal Muscle Phosphoproteome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Stuart Phillips, Professor, McMaster University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2196
Record Dates: First submitted 2020-02-05; First posted 2020-02-11 (Actual); Results first posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Skeletal Muscle Protein Synthesis
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Aerobic and resistance exercise
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): All subjects will perform both aerobic and resistance exercise
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Aerobic exercise and resistance exercise

SUMMARY:
Generally, resistance exercise increases muscle mass and strength, and fatigue resistance. How resistance exercise achieves these adaptations remains understudied, but what is known is that skeletal muscle translates the physical and biochemical stresses of resistance exercise into morphological and metabolic adaptations. While resistance exercise activates signaling pathways (i.e., proteins) that increase the synthesis of specific proteins to cause adaptations, thousands of proteins are likely involved, and their interactions are complicated. The investigators aim to study these processes.

DETAILED DESCRIPTION:
Skeletal muscle is a highly plastic tissue, capable of adapting to changes in nutritional intake and contractile activity. For instance, resistance exercise results in a mild stimulation of rates of muscle protein breakdown (MPB) but a greater stimulation of the rates of muscle protein synthesis (MPS). When resistance exercise is performed prior to protein ingestion there is a synergistic combination of the two stimuli such that rates of MPS are stimulated over and above those of MPB. Thus, repeated bouts of resistance exercise, when coupled with protein ingestion, result in the accretion of skeletal muscle protein referred to as hypertrophy. Importantly, by changing the nature of the exercise stimulus, it is possible to redirect the focus of the type of skeletal muscle proteins that are being synthesized. For example, prolonged and repeated lower-load dynamic stimulation of skeletal muscle (i.e., endurance exercise training) results in an increase in the expression of mitochondrial genes, proteins, and ultimately enhanced mitochondrial content, leading to a shift towards an oxidative phenotype, and improved fatigue resistance. Resistance exercise training also stimulates the transcription of genes and accrual of new muscle proteins, but these genes and proteins are largely associated with the myofibrillar protein fraction, and regular resistance exercise leads to muscle hypertrophy and increased force-generating capacity. However, during the early stages of exercise training, particularly in training-naïve participants there is a significant increase in the expression of genes common to both modalities of exercise. It is only with sustained exercise training that there is a 'fine-tuning' of the transcriptome, the protein synthetic response, and then the proteome that gives rise to divergent hypertrophic and oxidative phenotypes.

ELIGIBILITY:
Inclusion Criteria:

- between the ages of 18 and 30 years

Exclusion Criteria:

* Smoker or user of tobacco products;
* High physical activity
* Have health problems such as: renal or gastrointestinal disorders, metabolic disease, heart disease, vascular disease, rheumatoid arthritis, diabetes, poor lung function, uncontrolled blood pressure, dizziness, thyroid problems, or any other health conditions for which you are being treated that might put you at risk for this study;
* Taking anti-diabetic, anti-inflammatory, platelet inhibitor, or anti-coagulant medications;
* Use of an investigational drug product within the last 30 days;
* Have participated in an infusion protocol in the last year; or
* Do not understand English or have a condition the PI believes would interfere with a participants' ability to provide informed consent, comply with the study protocol, or which might confound the interpretation of the study results or put someone at undue risk.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2024-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Phillips, PhD, Principal Investigator — McMaster University, Department of Kinesiology
Locations (1):
- Exercise Metabolism Research Laboratory, McMaster Univeristy, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All data will be deposited on OSF
Supporting Information: Study Protocol, CSR
Time Frame: At the time of publication
Access Criteria: Everyone can access

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exercise
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Exercise
Number analyzed (Participants) | 16
Age, Customized [Mean (Full Range); unit: Years]
  Age | 21 [19 to 26]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Muscle Protein Synthesis [Mean (Standard Deviation); unit: Protein synthesis (% / hour)] — Myofibrillar MPS will be calculated using the precursor-product equation: myofibrillar MPS = ([E2b-E1b]/[Eic x t]) x 100. Eb represents the enrichment of bound myofibrillar protein, Eic is the average intracellular enrichment between two biopsies, and t is the tracer incorporation time in hours. Final units expressed as a relative rate of synthesis (% per hour).
  As we will employ 'tracer naïve' participants (had not previously participated in a study protocol where L-[ring- 13C6] phenylalanine was infused), a pre-infusion blood sample will be used for the calculation of resting MPS. Population: Two cohorts recruited and analyzed separately.
  Protein synthesis (% / hour)
    Cohort 1: number analyzed (Participants) | 4
    Cohort 1 | 0.041 (0.007)
    Cohort 2: number analyzed (Participants) | 12
    Cohort 2 | 0.027 (0.004)

OUTCOME MEASURES:

1. Primary Outcome: Change in Acute Muscle Protein Synthesis
Description: Myofibrillar and intracellular enrichments of L-[ring- 13C6] phenylalanine will be measured. MPS will be calculated using the precursor-product equation: MPS =([E2b-E1b]/[Eic x t]) x 100. Eb represents the enrichment of bound myofibrillar protein, Eic is the average intracellular enrichment between two biopsies, and t is the tracer incorporation time in h. As we will employ 'tracer naïve' participants (had not previously participated in a study protocol where L-[ring- 13C6] phenylalanine was infused), a pre-infusion blood sample will be used for the calculation of resting myofibrillar MPS. The outcomes measure will be expressed as a percentage change of MPS relative to the baseline measure. i.e. intracellular enrichment of L-[ring- 13C6] phenylalanine relative to the baseline (resting) period.
Time Frame: Pre exercise (resting) to 3 hours post-exercise
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Exercise
Number analyzed (Participants) | 12
percent change
  Myofibrillar Protein Synthesis | 143 (53)
  Sarcoplasmic Protein Synthesis | 123 (115)

ADVERSE EVENTS:
Time Frame: Data for adverse events were collected over a period of 6 weeks.
Arm/Group | Exercise
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-05): https://cdn.clinicaltrials.gov/large-docs/14/NCT04263714/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-05): https://cdn.clinicaltrials.gov/large-docs/14/NCT04263714/ICF_001.pdf